CLINICAL TRIAL: NCT04903938
Title: Primary And Secondary Abilities Among The Individuals With Antisocial Personality Disorder Within The Scope Of Positive Psychotherapy: Their Relationship With Criminal Behaviors, Aggression And Anger.
Brief Title: Positive Psychotheraphy and Antisocial Personality Disorder: Crime, Aggression, Anger
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: Sultan Abdulhamid Han TaRH
Record Dates: First submitted 2021-05-15; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Antisocial Personality Disorder
Keywords: Antisocial personality disorder; Primary abilities; Secondary abilities; Positive psychotheraphy; Anger; Aggression
MeSH Terms: conditions — Antisocial Personality Disorder; Aggression | interventions — mycophenolic adenine dinucleotide; Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Criminal-Antisocial Personality Disorder: The study groups were determined as those with criminal antisocial personality disorder, those with non-criminal antisocial personality disorder and the control group. Those with antisocial personality disorder were divided into criminal and non-criminal groups according to their criminal records. The number of groups was determined as three with the control group.
  Interventions: Behavioral: Primary And Secondary Abilities Among The Individuals With Antisocial Personality Disorder Within The Scope Of Positive Psychotherapy: Their Relationship With Criminal Behaviors, Aggression And Anger
- Non-criminal group: The study groups were determined as those with criminal antisocial personality disorder, those with non-criminal antisocial personality disorder and the control group. Those with antisocial personality disorder were divided into criminal and non-criminal groups according to their criminal records. The number of groups was determined as three with the control group.
  Interventions: Behavioral: Primary And Secondary Abilities Among The Individuals With Antisocial Personality Disorder Within The Scope Of Positive Psychotherapy: Their Relationship With Criminal Behaviors, Aggression And Anger
- Control group: The study groups were determined as those with criminal antisocial personality disorder, those with non-criminal antisocial personality disorder and the control group. Those with antisocial personality disorder were divided into criminal and non-criminal groups according to their criminal records. The number of groups was determined as three with the control group.
  Interventions: Behavioral: Primary And Secondary Abilities Among The Individuals With Antisocial Personality Disorder Within The Scope Of Positive Psychotherapy: Their Relationship With Criminal Behaviors, Aggression And Anger

INTERVENTIONS:
Behavioral: Primary And Secondary Abilities Among The Individuals With Antisocial Personality Disorder Within The Scope Of Positive Psychotherapy: Their Relationship With Criminal Behaviors, Aggression And Anger — Participants will be given scales with validity and reliability studies in Turkish.
  Other Names: Investigation of primary and secondary abilities, criminal behavior, aggression and anger behaviors in patients with criminal antisocial personality disorder and comparison with other's data; Investigation of primary and secondary abilities, criminal behavior, aggression and anger behaviors in patients with non-criminal antisocial personality disorder and comparison with other's data; Investigation of primary and secondary abilities, criminal behavior, aggression and anger behaviors in patients with control group and comparison with other's data

SUMMARY:
Studies on Antisocial Personality Disorder (ASPD), in which criminal behaviors, aggression and anger behaviors are frequently seen, are very rare. Developed by Nosrat Peseschkian, positive psychotherapy is an eclectic therapy approach born from the psychodynamic approach, existential-humanist approach, behavioral approach and intercultural therapy approach. Psychodynamic psychotherapy is a humanistic, psychodynamic, resource-focused, conflict-solving, integrative and intercultural approach that has its own unique intervention methods as well as the features of other therapy theories. In this study, it was aimed to determine the primary and secondary abilities of individuals with criminal and non-criminal antisocial personality disorder within the scope of positive psychotherapy, to compare these abilities with respect to healthy individuals, and to examine the effects on crime, aggression behavior and anger levels.

DETAILED DESCRIPTION:
Antisocial personality disorder usually begins before the age of 15 and is characterized by neglect and violation of the rights of others, impulsivity, aggression, apathy, irresponsibility, and criminal behavior. Lack of empathy, anger, anger and hostility, and confrontation with legal problems can be seen in those with antisocial personality disorder.

Epidemiological studies of antisocial personality disorder are scarce and focus predominantly on all adults, especially young adults. The frequency of ASPD among adults in the general population is estimated at 3.0% - 4.3%. Antisocial personality disorder is 3.5 times more common in men than in women. Genetic and environmental factors play a role in the etiology of this disorder. In addition, mental disorders such as major depressive disorder, generalized anxiety disorder and substance use disorders are frequently encountered in these individuals.

Individuals with antisocial personality disorder often exhibit aggressive behavior. Aggressive behaviors have been associated with risk factors such as low household income, insufficient parental control, single-parent families, upbringing by antisocial parents, neglect, and presence of criminal peer relationships. Modeling of aggressive behaviors can be explained as part of the individual's problems related to the environment in which he grows and his attachments, and by taking the aggressive behaviors witnessed as an example.

The positive concept is derived from the expression "positum" and means existing, real, actual, given, real and concrete. This concept reflects the focus of the positive psychotherapy approach because the method motivates the client's capacities to find out what the symptom is doing to resolve the conflict and find a useful solution.

Positive psychotherapy is an eclectic approach stemming from psychodynamic approach, existential-humanistic approach, behavioral approach and intercultural therapy approach. In addition, positive psychotherapy is a humanistic, psychodynamic, resource-focused, conflict-solving, complementary and intercultural approach that incorporates features of other therapy-related theories as well as original intervention procedures. While this theory, like other therapy theories, aims to treat disorders and diseases, it places special emphasis on one's abilities and development possibilities. According to the positive psychotherapy approach, although each person has such abilities, the intensity is different. In this sense, although it is important in a positive psychotherapy approach to accept problems and disorders as they are, it is also important to focus on things outside of them, take into account any person's current abilities, and help clients realize their abilities and capacities. Almost all consulting approaches can focus on this point. However, unlike other approaches, the positive psychotherapy approach places a central emphasis on this issue and puts it into practice within a meta-theory for the treatment plan.

The principles of balance, consultation and hope are the three basic principles of positive psychotherapy. If the client continues to live a balanced life in key areas such as body, success, contact and future / fantasy / spirituality, they gain a balance model. The principle of consultation means that the client cooperates with the individuals around him to solve his problems. The hope principle is that the client believes that they can solve their problems and overcome them.

Positive psychotherapy approach argues that people come to the world with two important abilities: the ability to love and the ability to know. The ability to know manifests itself in secondary abilities. Patience, time, love, trust, faith, hope, contact and tenderness / sexuality are evaluated within the primary abilities. Secondary abilities include order, cleanliness, punctuality, politeness, honesty, archievement, reliability, thrift, obedience, justice and faitfulness. This type of therapy conception links the emergence of mental disorders to the underdevelopment or overdevelopment of these abilities. The positive psychotherapy approach focuses on the optimal use of these abilities.

Structured cognitive behavioral techniques, psychoanalytic psychotherapy, dialectical behavior therapy, schema-focused therapy, and mindfulness-based therapy are used to treat antisocial personality disorder. In addition to these intervention methods, positive psychotherapy discusses the hypothetical statements regarding antisocial personality disorder.

Positive psychotherapy explains that personality development takes place through abilities. It is an important assumption that many skills suggested by this approach predict aggression and anger levels in cases with antisocial personality disorder. Studies on aggression, anger, and delinquent behaviors in studies conducted with individuals with Antisocial Personality Disorder are available in the literature. However, there are no studies addressing these behaviors within the scope of positive psychotherapy.

According to the researchers' knowledge, this study is the first study to examine the primary and secondary abilities of individuals with criminal and non-criminal antisocial personality disorder within the scope of positive psychotherapy and the effect of these abilities on criminal behavior and aggression and anger levels.

It is thought that determining the abilities of individuals with criminal and non-criminal antisocial personality disorder within the scope of positive psychotherapy and explaining the behavioral pathologies in these individuals will contribute to the literature. In this context, the purpose of this study is to compare the primary and secondary abilities of individuals with antisocial personality disorder within the scope of positive psychotherapy with healthy individuals and to examine whether these abilities are associated with criminal behavior, anger and aggression tendencies in individuals with antisocial personality disorder. In addition, it is to bring a new perspective to the studies of those with antisocial personality disorder and to provide a perspective for future studies. The findings of this study can be used by therapists working with individuals with criminal and non-criminal antisocial personality disorder in the process of positive psychotherapy and may eliminate the gap in this area.

Before starting the study, approval was obtained from the local ethics committee. Including individuals who were older than 18 years of age, who were able to read and understand structured interview forms and scale forms, and who were at the education level (at least primary school graduate), who agreed to participate in the study, and who were diagnosed with Antisocial Personality Disorder according to SCID-1 and DSM IV diagnostic criteria. has been. Those under the age of 18, those who did not agree to participate in the study, those with a comorbid psychiatric disorder according to SCID-1 and DSM IV diagnostic criteria, and those with an additional medical disease were excluded from the study. The researchers interviewed the participants face to face and provided information about the study. Participants were given a structured interview form prepared by the researchers, the Wiesbaden Positive Psychotherapy and Family Therapy Inventory that evaluates primary and secondary abilities, the Buss-Perry Impulsivity Scale to determine the levels of aggression, and the Trait Anger and Anger Expression Scale to determine the levels of anger. The data of the study were obtained in this way.

Statistical analysis of the study data was made using the SPSS 15.0 package program. Number, percentage, average and standard deviation values will be used in defining the data. Student T test will be used for continuous variables in comparisons between groups, and Chi-Square test will be used for comparing discrete variables. Pearson correlation analysis will be used to examine the relationships between variables. A level of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Be over 18 years of age,
2. To be at an educational level that can take tests and structured interview form (at least primary school graduate)
3. To agree to participate in the study, D. Being diagnosed with Antisocial Personality Disorder according to SCID-2 and DSM IV diagnostic criteria, to. Alcohol-Substance abuse and / or dependence,

Exclusion Criteria:

1. Being under the age of 18,
2. Refusing to participate in the study,
3. Having a comorbid psychiatric disorder according to SCID-1 and DSM IV diagnostic criteria,
4. Having an additional medical disease, to. Alcohol-substance use and not being addicted,

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility of the participant is based on self-representation of gender identity.
Study Population: 100+100
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Primary and secondary abilities, aggression and anger levels of criminal antisocial personality disorder | September 2013
  Determination of primary and secondary abilities, aggression and anger levels of those with criminal antisocial personality disorder
The relationship between primary and secondary abilities and aggression and anger levels of criminal antisocial personality disorder | September 2013
  Determining the relationship between primary and secondary abilities and aggression and anger levels of those with criminal antisocial personality disorder
Primary and secondary abilities, aggression and anger levels of non-criminal antisocial personality disorder | September 2013
  Determination of primary and secondary abilities, aggression and anger levels of those with non-criminal antisocial personality disorder
The relationship between primary and secondary abilities and aggression and anger levels of non-criminal antisocial personality disorder | September 2013
  Determining the relationship between primary and secondary abilities and aggression and anger levels of those with non-criminal antisocial personality disorder
Primary and secondary abilities, aggression and anger levels of control group | September 2013
  Determining the relationship between primary and secondary abilities and aggression and anger levels of control group
Comparison of the primary and secondary abilities, aggression and anger levels of those with criminal antisocial personality disorder with those with non-criminal antisocial personality disorder and the control group | September 2013
  Comparison of the primary and secondary abilities, aggression and anger levels of those with criminal antisocial personality disorder with those with non-criminal antisocial personality disorder and the control group

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: june 2026

REFERENCES:
- [Background] Stoddard SA, Zimmerman MA, Bauermeister JA. Thinking about the future as a way to succeed in the present: a longitudinal study of future orientation and violent behaviors among African American youth. Am J Community Psychol. 2011 Dec;48(3-4):238-46. doi: 10.1007/s10464-010-9383-0. PMID 21104432
- [Result] Derefinko, K. J., & Widiger, T. A. (2016). Antisocial personality disorder. In: S. H. Fatemi & P. J. Clayton (Eds.), The medical basis of psychiatry, 4th edn. Springer, New York; 2016,229-245. https://doi.org/10.1007/978-1-4939-2528-5_13
- [Result] Volkert J, Gablonski TC, Rabung S. Prevalence of personality disorders in the general adult population in Western countries: systematic review and meta-analysis. Br J Psychiatry. 2018 Dec;213(6):709-715. doi: 10.1192/bjp.2018.202. Epub 2018 Sep 28. PMID 30261937
- [Result] Goldstein RB, Chou SP, Saha TD, Smith SM, Jung J, Zhang H, Pickering RP, Ruan WJ, Huang B, Grant BF. The Epidemiology of Antisocial Behavioral Syndromes in Adulthood: Results From the National Epidemiologic Survey on Alcohol and Related Conditions-III. J Clin Psychiatry. 2017 Jan;78(1):90-98. doi: 10.4088/JCP.15m10358. PMID 27035627
- [Result] Farrington, D. P., & Bergstrøm, H. (2018). Family background and psychopathy. In C. J. Patrick (Ed.), Handbook of psychopathy, 2nd Ed. (54-379). The Guilford Press.
- [Result] Eron, L. D. (1997). The development of antisocial behavior from a learning perspective. In D. M. Stoff, J. Breiling, & J. D. Maser (Eds.), Handbook of antisocial behavior (p. 140-147). John Wiley & Sons Inc.
- [Result] Sarı, T. (2015). Positive psychotherapy: Its development, basic principles and methods and applicability to Turkish culture. The Journal of Happiness Well-Being, 3, 182-203.
- [Result] Peseschkian, N., Walker, R. K. (2013). Positive Psychotherapy in Psychosomatic Medicine: A Transcultural and Interdisciplinary Approach: Examining 40 Disorders, Walker, R. K. (Translator Ed.), Wiesbaden, Germany.
- [Result] Peseschkian, N. (2015). Introduction to Positive Psychotherapy, Theory and Practice; Sarı T. (Trans. ed.), 1st Edition, Anı Press, Ankara.
- [Result] Sinici, E., Sarı, T., & Maden, Ö. (2014). Primary and secondary capacities of post-traumatic stress disorder patients in terms of positive psychotherapy. International Journal of Psychotherapy 18, 22-34.
- [Result] Sinici, E. (2017). Primary and Secondary Capacities of First Grade Nursing Students in the Context of Positive Psychotherapy. International Journal of Psychotherapy, January 21,1.
- [Result] Barbaree HE. Psychopathy, treatment behavior, and recidivism: an extended follow-up of Seto and Barbaree. J Interpers Violence. 2005 Sep;20(9):1115-31. doi: 10.1177/0886260505278262. PMID 16051730
- [Result] Loginov, S. A. (2017). Simlarities And Differences In Approaches Of Cognitive Therapy And Modern Psychoanalysis To Antisocial Personlity Disorder. Международный научно-исследовательский журнал, (02 (56) Часть 3), 63-65. https://doi.org/10.23670/IRJ.2017.56.085
- [Result] Neacsiu AD, Tkachuck MA. Dialectical behavior therapy skills use and emotion dysregulation in personality disorders and psychopathy: a community self-report study. Borderline Personal Disord Emot Dysregul. 2016 Jul 20;3:6. doi: 10.1186/s40479-016-0041-5. eCollection 2016. PMID 27446589
- [Result] Young, J. E., Klosko, J. S., & Weishaar, M. E. (2003). Schema therapy. New York: Guilford, 254.
- [Result] Stratton, K. J. (2006). Mindfulness-based approaches to impulsive behaviors. The New School Psychology Bulletin, 4(2), 49-71.
- [Result] First, M. B., Spitzer, R. L., Gibbon, M., & Williams, J. B. W. (1997). User's guide for the Structured Clinical Interview for DSM-IV Axis I Disorders. Washington, DC: American Psychiatric Press
- [Result] Corapcioglu A, Aydemir O, Yildiz M, Esen A, Koroglu E. (1999). Structured clinical interview for DSM-IV axis I disorders (SCID-I), clinical version. Ankara: Hekimler Yayin Birligi, 1999.
- [Result] Spitzer RL, Spitzer RL. (1989). Instruction manual for the Structured Clinical Interview for DSM-III-R (SCID). Biometrics Research Department, New York State Psychiatric Institute.
- [Result] Sorias, S., Saygılı, R., Elbi, H., Vahip, S., Mete, L., & Nifirne, Z. (1990). Structured clinical interview for DSM-III-R personality disorders, Turkish version. Izmir: Ege Universitesi Basimevi.
- [Result] Peseschkian, N., & Deidenbach, H. (1988). Wiesbadener Inventar zur Positiven Psychotherapie und Familientherapie: WIPPF. Springer.
- [Result] Sarı, T., Eryılmaz, A., & Varlıklı-Öztürk, G. (2010). Adaption of Wiesbaden inventory of positive psychotherapy to Turkish culture. Oral Present 5th World Congr Posit Psychother, 9-
- [Result] Spielberger, C. D., Jacobs, G., Russell, S., & Crane, R. S. (1983). Assessment of anger: The state-trait anger scale. Advances in personality assessment, 2, 161-189.
- [Result] Ozer, A. K. (1994). Continuous Anger and Anger Expression Style Preliminary Study. Turkish Journal of Psychology, 9(31), 26-35.
- [Result] Buss AH, Perry M. The aggression questionnaire. J Pers Soc Psychol. 1992 Sep;63(3):452-9. doi: 10.1037//0022-3514.63.3.452. PMID 1403624
- [Result] Demirtas Madran HA. [The reliability and validity of the Buss-Perry Aggression Questionnaire (BAQ)-Turkish Version]. Turk Psikiyatri Derg. 2013 Summer;24(2):124-9. Turkish. PMID 23754266
- [Result] Peseschkian, N. (2002). Günlük yaşamın psikoterapisi (Çev. H. Fışıloğlu). Istanbul: Beyaz Press.
- [Result] Kızmaz, Z. (2005). An evaluation on the potential of sociological crime theories to explain the phenomenon of crime. Cumhuriyet University Journal of Social Sciences, 29(2):149-74.
- [Result] Agnew, R. (2001). Building on the foundation of general strain theory: Specifying the types of strain most likely to lead to crime and delinquency. Journal of research in crime and delinquency, 38(4), 319-361. https://doi.org/10.1177/0022427801038004001
- [Result] Correa-Chávez, M., Mejía-Arauz, R., & Rogoff, B. (2015). Children learn by observing and contributing to family and community endeavors: A cultural paradigm. Academic Press.
- [Result] Baker, L., Jaffe, P., & Moore, K. (2001). Understanding the effects of domestic violence: A trainer's manual for early childhood educators. London, ON: Centre for Children & Families in the Justice System.
- [Result] Hegarty K, Taft A, Feder G. Violence between intimate partners: working with the whole family. BMJ. 2008 Aug 4;337:a839. doi: 10.1136/bmj.a839. No abstract available. PMID 18678595
- [Result] Clarke, J. (2009). Working With Monsters: How to Identify and Protect Yourself from the Workplace Psychopath: Easyread Super Large 20pt Edition. ReadHowYouWant. com.
- [Result] Reeves, M., & Taylor, J. (2007). Specific relationships between core beliefs and personality disorder symptoms in a non-clinical sample. Clinical Psychology & Psychotherapy: An International Journal of Theory & Practice, 14(2), 96-104. https://doi.org/10.1002/cpp.519
- [Result] Ovacık, A.C. (2008). The effects of domestic violence on male child's violent criminal behavior. Master Thesis, Istanbul University Institute of Forensic Medicine, Istanbul.